CLINICAL TRIAL: NCT04791085
Title: Investigation of Stress Levels and Lifestyle of a Sample of Greek General Surgeons in Covid-19 and Non-reference Hospitals
Brief Title: Investigation of Stress Levels and Lifestyle of a Sample of Greek General Surgeons in Covid-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Amalia Fleming General Hospital (Other)
Responsible Party: Principal Investigator, Petros Loukas Chalkias, Principal Investigator, National and Kapodistrian University of Athens
Other Study IDs: 1183/17.02.21
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Stress, Psychological; Stress, Emotional; Life Style Induced Illness; Anxiety Depression; Covid19
MeSH Terms: conditions — Stress, Psychological; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- general surgeons: General surgeons who work at general or private hospitals in Greece

SUMMARY:
A new pandemic appeared in early 2020, also known as the coronavirus (Covid-19), affecting all health systems worldwide. Medical and nursing staff make every effort to treat patients resulting in physical and psychological exhaustion, which is exacerbated by the lack of medical and nursing staff, the lack of protective equipment, the increased workload, and increased shifts.

In this context, the surgeons had to contribute in turn, in order to help as much as they could in dealing with this new health crisis, as a result of which they find themselves in positions that are not on their subject or in their proper training and to handle patients with a dangerous and highly aggressive respiratory infection. This brought more psychological and physical stress to the surgeons. The pandemic of Covid-19 is not known to be a purely surgical condition, but many patients with coronavirus require surgery due to an additional infection, condition, or complication.

The design of this research will be observational and quantitative. Quantitative design involves the provision of numerically coded and analytical measurements, such as self-report questionnaires.

The purpose of this cross-sectional research is primarily to record the levels of stress, anxiety, depressive symptoms of Greek surgeons, and their lifestyle. Secondary to correlate the stress levels with socio-demographic data and their lifestyle with other parameters of the study.

DETAILED DESCRIPTION:
A new pandemic emerged in early 2020, also known as the coronavirus (Covid-19) pandemic, affecting all health systems worldwide. This disease, although it attacks the human respiratory system, has greatly affected all health personnel regardless of specialty and the reason is that these patients need a high level of care. Medical and nursing staff make every effort to treat patients resulting in physical and psychological exhaustion, which is exacerbated by the lack of medical and nursing staff, the lack of protective equipment, the increased workload. and increased shifts.

In this context, the surgeons had to contribute in turn, in order to help as much as they could in dealing with this new health crisis, as a result of which they find themselves in positions that are not on their subject or in their proper training and to handle patients with a dangerous and highly aggressive respiratory infection. This brought more psychological and physical stress to the surgeons.

Their presence in aerosol situations (surgeries - intubation, placement of central venous catheters) and frequent contact with patients increased the likelihood of disease spread. With the increased likelihood of the disease spreading as their exposure to patients was high, it began to cause concern to staff living with the elderly or other vulnerable groups.

The incidence of the Covid-19 pandemic is increasing rapidly, resulting in worldwide healthcare systems operating feverishly to adequately meet the demands of this new disease. Several countries around the world have converted general hospitals to host hospitals exclusively for this disease, as a safety measure and limitation of the spread of Covid-19.

Front-line health personnel is under stress due to increased workload, lack of protective equipment, lack of information, and social isolation from loved ones. This staff includes physicians, pulmonologists, intensivists, surgeons.

In the last decade, there has been a great deal of mobility in the health sciences with reference to stress as many studies have linked it to the occurrence of various physical and psychological disorders. Undoubtedly, stress is a multifactorial concept, which makes it difficult to define clearly.

Stress, in particular, is a response mechanism, a "fight or flight" reflex in order to protect the body from various dangers. It is always activated with the "perception" of danger or threat (real or imaginary), where the sympathetic fate of the autonomic nervous system is stimulated and aims to prepare the body either to escape from danger or to fight with it.

The stressors that affect surgeons are many and varied, such as minimal sleep and its disturbance with multiple shifts, workplace tension, heavy workload, poor diet, etc. Depending on the stressors, the stress axis is activated with the corresponding effects on their psychosomatic health (depression, burnout, obesity, cardiovascular and autoimmune diseases).

Based on the above, the present study has not so far looked more broadly at the psychological stress of surgeons in relation to their quality of life during the Covid-19 period.

The design of this research will be observational and quantitative. Quantitative design involves the provision of numerically coded and analytical measurements, such as self-report questionnaires (social-demographic data, DASS-21, Anxiety Covid-19, Pittsburgh, Healthy Lifestyle and Personal Control Questionnaire, Multidimensional Health Locus of Control).

The purpose of this cross-sectional research is primarily to record the levels of stress, anxiety, depressive symptoms of Greek surgeons, and their lifestyle. Secondary to correlate the stress levels with socio-demographic data and their lifestyle with other parameters of the study.

ELIGIBILITY:
Inclusion Criteria:

* participants will be surgeons or interns of general surgery in any hospital in Greece.

Exclusion Criteria:

* participants who will practice another medical specialty

Ages: 23 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Greek general surgeons and interns of general surgery working in private and general hospitals in the country.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-05-08 (Estimated); Study Completion 2021-05-08 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | day 1
  most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress.PSS scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the four positively stated items (items 4, 5, 7, & 8) and then summing across all scale items. A short 4 item scale can be made from questions 2, 4, 5 and 10 of the PSS 10 item scale.
DASS-21 | day 1
  The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items.Recommended cut-off scores for conventional severity labels (normal, moderate, severe) are as follows:Depression normal 0-9, mild 10-13, moderate 14-20, severe 21-27, extremely severe 28+, Anxiety normal 0-7, mild 8-9, moderate 10-14, severe 15-19, extremely severe 20+, Stress normal 0-14, mild 15-18, moderate 19-25, severe 26-33, extremely severe 34+
PITTSBURGH (GR-PSQI) | day 1
  The PSQI includes a scoring key for calculating a patient's seven subscores, each of which can range from 0 to 3. The subscores are tallied, yielding a "global" score that can range from 0 to 21. A global score of 5 or more indicates poor sleep quality; the higher the score, the worse the quality.
Healthy Lifestyle and Personal Control Questionnaire | day 1
  the Healthy Lifestyle and Personal Control Questionnaire (HLPCQ),which aims to assess the concept of empowerment through a constellation of daily activities.1) Dietary Healthy Choices, 2) Dietary Harm Avoidance, 3) Daily Routine, 4) Organized Physical Exercise and 5) Social and Mental Balance. All subscales showed satisfactory internal consistency and variance, relative to theoretical score ranges. Subscale scores and the total score were significantly correlated with perceived stress and health locus of control, implying good criterion validity. Associations with sociodemographic data and other variables, such as sleep quality and health assessments, were also found.The HLPCQ is a good tool for assessing the efficacy of future health-promoting interventions to improve individuals' lifestyle and wellbeing.
Multi dimensional Health Locus of Control (MHLC) | day 1
  The health control center will be evaluated using the Multi dimensional Health Locus of Control (MHLC). The MHLC consists of three sub-scales that assess whether the respondent attributes the outcome of his or her health events to luck, to himself or to others. This questionnaire consists of a total of 18 questions with possible answers from ("I strongly disagree") to 6 ("I strongly agree"). For each sub-scale, high values mean strong performance on this factor.
COVID-19-Anxiety Questionnaire (C-19-A) | day 1
  Participants' concerns about covid-19 will be measured using the COVID-19-Anxiety Questionnaire (C-19-A). This measurement tool consists of 10 questions that are scored on a Likert scale with values from 0 (not at all) to 4 (too much). High prices reflect high concern.

CONTACTS AND LOCATIONS:
Overall Officials: Petros L Chalkias, MD, Principal Investigator — Sismanoglio - Amalia Fleming General Hospital
Locations (1):
- Sismanoglio-Amalia Fleming Hospital, Athens, Melissia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nickell LA, Crighton EJ, Tracy CS, Al-Enazy H, Bolaji Y, Hanjrah S, Hussain A, Makhlouf S, Upshur RE. Psychosocial effects of SARS on hospital staff: survey of a large tertiary care institution. CMAJ. 2004 Mar 2;170(5):793-8. doi: 10.1503/cmaj.1031077. PMID 14993174
- [Background] Chan AO, Huak CY. Psychological impact of the 2003 severe acute respiratory syndrome outbreak on health care workers in a medium size regional general hospital in Singapore. Occup Med (Lond). 2004 May;54(3):190-6. doi: 10.1093/occmed/kqh027. PMID 15133143
- [Background] Rossi R, Socci V, Pacitti F, Di Lorenzo G, Di Marco A, Siracusano A, Rossi A. Mental Health Outcomes Among Frontline and Second-Line Health Care Workers During the Coronavirus Disease 2019 (COVID-19) Pandemic in Italy. JAMA Netw Open. 2020 May 1;3(5):e2010185. doi: 10.1001/jamanetworkopen.2020.10185. PMID 32463467
- [Background] Lai J, Ma S, Wang Y, Cai Z, Hu J, Wei N, Wu J, Du H, Chen T, Li R, Tan H, Kang L, Yao L, Huang M, Wang H, Wang G, Liu Z, Hu S. Factors Associated With Mental Health Outcomes Among Health Care Workers Exposed to Coronavirus Disease 2019. JAMA Netw Open. 2020 Mar 2;3(3):e203976. doi: 10.1001/jamanetworkopen.2020.3976. PMID 32202646
- [Background] Shanafelt T, Ripp J, Trockel M. Understanding and Addressing Sources of Anxiety Among Health Care Professionals During the COVID-19 Pandemic. JAMA. 2020 Jun 2;323(21):2133-2134. doi: 10.1001/jama.2020.5893. No abstract available. PMID 32259193
- [Background] Balibrea JM, Badia JM, Rubio Perez I, Martin Antona E, Alvarez Pena E, Garcia Botella S, Alvarez Gallego M, Martin Perez E, Martinez Cortijo S, Pascual Miguelanez I, Perez Diaz L, Ramos Rodriguez JL, Espin Basany E, Sanchez Santos R, Soria Aledo V, Lopez Barrachina R, Morales-Conde S. Surgical Management of Patients With COVID-19 Infection. Recommendations of the Spanish Association of Surgeons. Cir Esp (Engl Ed). 2020 May;98(5):251-259. doi: 10.1016/j.ciresp.2020.03.001. Epub 2020 Apr 3. PMID 32252979
- [Background] Brat GA, Hersey S, Chhabra K, Gupta A, Scott J. Protecting Surgical Teams During the COVID-19 Outbreak: A Narrative Review and Clinical Considerations. Ann Surg. 2023 Nov 1;278(5):e957-e959. doi: 10.1097/SLA.0000000000003926. Epub 2020 Apr 17. No abstract available. PMID 32379080